CLINICAL TRIAL: NCT00050622
Title: ADHD Treatment: Comparative and Combined Dosage Effects
Brief Title: Behavioral Treatment, Drug Treatment, and Combined Treatment for Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: R01MH062946 (NIH); R01MH062946 (NIH); DSIR CT-CT
Record Dates: First submitted 2002-12-16; First posted 2002-12-17 (Estimated); Results first posted 2016-09-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (12):
- No Treatment (Placebo Comparator): No Medication, No Behavior Modification (BMOD)
  Interventions: Drug: Placebo
- Low Dose Medication Only (Active Comparator): 0.15 mg/kg methylphenidate (MPH), No BMOD
  Interventions: Drug: Methylphenidate 0.15 mg/kg
- Medium Dose Medication Only (Active Comparator): 0.3 mg/kg MPH, No BMOD
  Interventions: Drug: Methylphenidate 0.3 mg/kg
- Higher Dose Medication Only (Active Comparator): 0.6 mg/kg MPH, No BMOD
  Interventions: Drug: Methylphenidate 0.6 mg/kg
- Low Intensity BMOD Only (Active Comparator): Placebo, Low Intensity BMOD
  Interventions: Behavioral: Low-Intensity BMOD; Drug: Placebo
- Low Intensity BMOD + Low Dose Medication (Active Comparator): 0.15 mg/kg MPH, Low Intensity BMOD
  Interventions: Drug: Methylphenidate 0.15 mg/kg; Behavioral: Low-Intensity BMOD
- Low Intensity BMOD + Medium Dose Medication (Active Comparator): 0.3 mg/kg MPH, Low Intensity BMOD
  Interventions: Behavioral: Low-Intensity BMOD; Drug: Methylphenidate 0.3 mg/kg
- Low Intensity BMOD + Higher Dose Medication (Active Comparator): 0.6 mg/kg MPH, Low Intensity BMOD
  Interventions: Behavioral: Low-Intensity BMOD; Drug: Methylphenidate 0.6 mg/kg
- High Intensity BMOD Only (Active Comparator): Placebo, High Intensity BMOD
  Interventions: Behavioral: High Intensity BMOD
- High Intensity BMOD + Low Dose Medication (Active Comparator): 0.15 mg/kg MPH, High Intensity BMOD
  Interventions: Drug: Methylphenidate 0.15 mg/kg; Behavioral: High Intensity BMOD
- High Intensity BMOD + Medium Dose Medication (Active Comparator): 0.3 mg/kg MPH, High Intensity BMOD
  Interventions: Drug: Methylphenidate 0.3 mg/kg; Behavioral: High Intensity BMOD
- High Intensity BMOD + Higher Dose Medication (Active Comparator): 0.6 mg/kg MPH, High Intensity BMOD
  Interventions: Drug: Methylphenidate 0.6 mg/kg; Behavioral: High Intensity BMOD

INTERVENTIONS:
Drug: Methylphenidate 0.15 mg/kg — 0.15 m/kg/dose immediate-release methylphenidate
  Arms: High Intensity BMOD + Low Dose Medication; Low Dose Medication Only; Low Intensity BMOD + Low Dose Medication
Behavioral: Low-Intensity BMOD — Lower-intensity behavioral treatment package.
  Arms: Low Intensity BMOD + Higher Dose Medication; Low Intensity BMOD + Low Dose Medication; Low Intensity BMOD + Medium Dose Medication; Low Intensity BMOD Only
Drug: Methylphenidate 0.3 mg/kg — 0.3 mg/kg/dose immediate-release methylphenidate
  Arms: High Intensity BMOD + Medium Dose Medication; Low Intensity BMOD + Medium Dose Medication; Medium Dose Medication Only
Drug: Placebo
  Arms: Low Intensity BMOD Only; No Treatment
Drug: Methylphenidate 0.6 mg/kg — 0.3 mg/kg/dose immediate-release methylphenidate
  Arms: High Intensity BMOD + Higher Dose Medication; Higher Dose Medication Only; Low Intensity BMOD + Higher Dose Medication
Behavioral: High Intensity BMOD — Comprehensive high-intensity Summer Treatment Program (STP)
  Arms: High Intensity BMOD + Higher Dose Medication; High Intensity BMOD + Low Dose Medication; High Intensity BMOD + Medium Dose Medication; High Intensity BMOD Only

SUMMARY:
The purpose of this study is to determine the effectiveness of behavioral treatment, drug treatment, and combined treatment for children with Attention Deficit Hyperactivity Disorder (ADHD). This study will also examine the interactions between different levels of behavioral and drug treatments.

DETAILED DESCRIPTION:
Participants attend a summer treatment program each Monday-Friday for 9 weeks. They participate in group recreational and classroom activities, with 12 children and 5 staff per group. Three behavioral conditions (no behavioral modification, low-intensity behavioral modification, and high-intensity behavioral modification) are delivered in random order, with each condition lasting 3 weeks. Along with the behavioral treatment conditions, children receive 1 of 4 medication doses (placebo, 0.15 mg/kg methylphenidate, 0.3 mg/kg methylphenidate, or 0.6 mg/kg methylphenidate) in random order, with each dose varied daily and repeated 3 or 4 times within each behavioral treatment condition.

Measures include frequency counts of positive and negative behaviors, academic productivity and accuracy in the classroom, and counselor, parent, and teacher ratings of benefits and side effects. Parents attend training sessions and implement behavioral programs at home.

ELIGIBILITY:
Inclusion Criteria:

* Attention Deficit Hyperactivity Disorder
* IQ >= 80

Exclusion Criteria:

* History of seizures or other neurological problems
* Medical history that would involve considerable risk in taking stimulant medication
* History or concurrent diagnosis of any of the following disorders: pervasive developmental disorder, schizophrenia or other psychotic disorders, sexual disorder, organic mental disorder, or eating disorder

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2001-09; Primary Completion 2004-08 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William E Pelham, PhD, Principal Investigator — Professor, Florida International University
Locations (2):
- United States (2):
  - Florida International University Center for Children and Families, Miami, Florida
  - Center for Children and Families, University at Buffalo, Buffalo, New York

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Fabiano, G.A., Pelham, W.E., Gnagy, E.M., Wymbs, B.T., Chacko, A., Coles, E.K., Walker, K.S., Arnold, F., Burrows-MacLean, L., Massetti, G.M., & Hoffman, M.T. (2007). The single and combined effects of multiple intensities of behavior modification and multiple intensities of methylphenidate in a classroom setting. School Psychology Review, 36(2), 195-216.
- [Background] Pelham WE, Burrows-MacLean L, Gnagy EM, Fabiano GA, Coles EK, Wymbs BT, Chacko A, Walker KS, Wymbs F, Garefino A, Hoffman MT, Waxmonsky JG, Waschbusch DA. A dose-ranging study of behavioral and pharmacological treatment in social settings for children with ADHD. J Abnorm Child Psychol. 2014 Aug;42(6):1019-31. doi: 10.1007/s10802-013-9843-8. PMID 24429997
- See also: Center for Children and Families Home Page — http://ccf.fiu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Within-Subject Treatment: All subjects received a within-subjects crossover of 3 levels of behavior modification, randomized in 3-week units, and 4 levels of medication, randomized on a daily basis. Thus each participant experienced all 12 combinations of No, Low, and High Intensity BMOD crossed with Placebo, 0.15 mg/kg MPH, 0.3 mg/kg MPH, and 0.6 mg/kg MPH conditions, with specific conditions changing daily.
Period: Overall Study
Arm/Group | Within-Subject Treatment
Started | 154
Completed | 153
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Within-Subject Treatment: All subjects completed a within-subjects crossover of 3 levels of behavior modification and 4 levels of medication.
Arm/Group | Within-Subject Treatment
Number analyzed (Participants) | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 154
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.15 (2.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 130
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 122
  More than one race | 9
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 154

OUTCOME MEASURES:

1. Primary Outcome: Social Behavior-Negative Verbalizations
Description: Sum of daily frequency of Verbal Abuse toward staff members, Teasing toward peers, and Cursing/Swearing as defined by a behavioral point system that doubles as an objective measure of children's behavior. All instances of these behaviors were reported and noted as they occur throughout daily activities.
Time Frame: Daily for 45 days
Measure: Mean (Standard Deviation); unit: Number of Observed Behaviors
Groups:
- No Treatment: No Medication, No BMOD
  Placebo
- Low Dose Medication Only: 0.15 mg/kg MPH, No BMOD
  Methylphenidate 0.15 mg/kg: 0.15 m/kg/dose immediate-release methylphenidate
- Low Intensity BMOD Only: Placebo, Low Intensity BMOD
  Low-Intensity BMOD: Lower-intensity behavioral treatment package.
  Placebo
- High Intensity BMOD Only: Placebo, High Intensity BMOD
  High Intensity BMOD: Comprehensive high-intensity STP
- High Intensity BMOD + Low Dose Medication: 0.15 mg/kg MPH, High Intensity BMOD
  Methylphenidate 0.15 mg/kg: 0.15 m/kg/dose immediate-release methylphenidate
  High Intensity BMOD: Comprehensive high-intensity STP
- High Intensity BMOD + Medium Dose Medication: 0.3 mg/kg MPH, High Intensity BMOD
  Methylphenidate 0.3 mg/kg: 0.3 mg/kg/dose immediate-release methylphenidate
  High Intensity BMOD: Comprehensive high-intensity STP
- High Intensity BMOD + Higher Dose Medication: 0.6 mg/kg MPH, High Intensity BMOD
  Methylphenidate 0.6 mg/kg: 0.3 mg/kg/dose immediate-release methylphenidate
  High Intensity BMOD: Comprehensive high-intensity STP
Arm/Group | No Treatment | Low Dose Medication Only | Medium Dose Medication Only | Higher Dose Medication Only | Low Intensity BMOD Only | Low Intensity BMOD + Low Dose Medication | Low Intensity BMOD + Medium Dose Medication | Low Intensity BMOD + Higher Dose Medication | High Intensity BMOD Only | High Intensity BMOD + Low Dose Medication | High Intensity BMOD + Medium Dose Medication | High Intensity BMOD + Higher Dose Medication
Number analyzed (Participants) | 153 | 153 | 153 | 153 | 153 | 153 | 153 | 153 | 153 | 153 | 153 | 153
Number of Observed Behaviors | 73.32 (127.11) | 45.41 (85.23) | 28.41 (59.11) | 15.08 (29.61) | 27.06 (45.77) | 13.70 (27.99) | 9.27 (20.05) | 4.28 (9.91) | 20.23 (41.13) | 7.61 (19.21) | 4.08 (8.59) | 2.49 (7.50)

2. Primary Outcome: Classroom Behavior
Description: Daily records of percentage of assigned problems completed by children in a 60-minute classroom period.
Time Frame: Daily for 45 days
Measure: Mean (Standard Deviation); unit: Percentage of Work Completed
Arm/Group | No Treatment | Low Dose Medication Only | Medium Dose Medication Only | Higher Dose Medication Only | Low Intensity BMOD Only | Low Intensity BMOD + Low Dose Medication | Low Intensity BMOD + Medium Dose Medication | Low Intensity BMOD + Higher Dose Medication | High Intensity BMOD Only | High Intensity BMOD + Low Dose Medication | High Intensity BMOD + Medium Dose Medication | High Intensity BMOD + Higher Dose Medication
Number analyzed (Participants) | 153 | 153 | 153 | 153 | 153 | 153 | 153 | 153 | 153 | 153 | 153 | 153
Percentage of Work Completed | 37 (23) | 53 (26) | 57 (24) | 61 (23) | 53 (21) | 67 (18) | 72 (19) | 75 (38) | 58 (22) | 72 (17) | 75 (14) | 76 (15)

3. Secondary Outcome: Treatment Satisfaction
Description: Parent rating of treatment satisfaction with medication, behavioral treatment, and their combination,on a scale of 1 (bad) to 7 (good).
Time Frame: End of Treatment
Measure: Mean (Standard Deviation); unit: Units on scale
Groups:
- No Treatment: No BMOD, No medication
- Medication Only: No BMOD + Medication (any dose)
- Low Intensity BMOD + Med: Low intensity behavior modification + medication (any dose)
- High Intensity BMOD + Medication: High Intensity BMOD + Medication (any dose)
Arm/Group | No Treatment | Low Intensity BMOD Only | High Intensity BMOD ONly | Medication Only | Low Intensity BMOD + Med | High Intensity BMOD + Medication
Number analyzed (Participants) | 143 | 143 | 143 | 143 | 143 | 143
Units on scale | 1.8 (1.2) | 2.7 (1.4) | 3.8 (1.6) | 3.5 (1.3) | 4.6 (1.3) | 5.6 (1.2)

ADVERSE EVENTS:
Time Frame: Daily for 45 days
Description: Parents completed the Pittsburgh Side Effects Rating Scale daily. Side effects were rated as None, Mild, Moderate, or Severe for common side effects of stimulant medication. Because the Side Effects Rating Scale applies only to medication side effects, treatment arms are collapsed across the three behavioral conditions.
Groups:
- Placebo: Placebo
- Low Dose Medication: 0.15 mg/kg MPH, No BMOD
- Medium Dose Medication: 0.3 mg/kg MPH, No BMOD
- Higher Dose Medication: 0.6 mg/kg MPH, No BMOD
Arm/Group | Placebo | Low Dose Medication | Medium Dose Medication | Higher Dose Medication
Serious Adverse Events (participants affected / at risk) | 0/154 | 0/154 | 0/154 | 0/154
Other Adverse Events (participants affected / at risk) | 3/153 | 2/153 | 3/153 | 17/153
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=153) | Low Dose Medication (N=153) | Medium Dose Medication (N=153) | Higher Dose Medication (N=153)
Tics (General disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) — Parent Rating of Moderate or Severe verbal or motor tics on the Pittsburgh Side Effects Rating Scale.
Picking at skin, nail biting (General disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) — Parent rating of Moderate or Severe on Pittsburgh Side Effects Rating Scale for picking at skin, nail biting, etc.
Buccal-Lingual Movements (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) — Parent rating of Moderate or Severe on Pittsburgh Side Effects Rating Scale for buccal-lingual movements
Worried/Anxious (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) — Parent rating of Moderate or Severe on Pittsburgh Side Effect Rating Scale for worry or anxiety
Dull, tired, listless (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Parent Rating of Moderate or Severe on Pittsburgh Side Effect Rating Scale for being dull, tired or listless.
Headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Parent Report of Moderate or Severe on Pittsburgh Side Effect Rating Scale for Headache.
Stomachache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Parent Rating of Moderate or Severe on Pittsburgh Side Effect Rating Scale for Stomach ache.
Irritability (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Parent Rating of Moderate or Severe on Pittsburgh Side Effects Rating Scale for Crabbiness/Irritability
Tearful, sad,depressed (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) — Parent Rating of Moderate or Severe on Pittsburgh Side Effects Rating Scale for tearfulness, sadness, or depression.
Social Withdrawal (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Parent Rating of Moderate or Severe on Pittsburgh Side Effects Rating Scale for social withdrawal
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Parent rating of Moderate or Severe on Pittsburgh Side Effects Rating Scale for hallucinations.
Trouble Sleeping (General disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (5) — Parent Rating of Moderate or Severe on Pittsburgh Side Effects Rating Scale for trouble sleeping.
Appetite Loss (General disorders) | 0 (0) | 1 (1) | 0 (0) | 9 (9) — Parent Rating of Moderate or Severe on Pittsburgh side Effects Rating Scale for appetite loss.

LIMITATIONS AND CAVEATS:
Highly structured environment and direct observational measures were used. Additional study in natural school and home settings will be necessary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes